CLINICAL TRIAL: NCT02551107
Title: Nasal Nitric Oxide Levels in Infants With and Without Congenital Heart Disease
Brief Title: Infant Nasal Nitric Oxide Levels in Congenital Heart Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate resources
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Principal Investigator, Lindsay Ryerson, Assistant Professor, University of Alberta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-LR-01
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Congenital heart disease (Experimental): Inclusion criteria: All participants, less than one year of age, with CHD will be eligible for this study with the exception of those patients with only patent foramen ovale (PFO) and patent ductus arteriosus (PDA). The diagnosis of CHD will be confirmed by echocardiography.
  Exclusion criteria: Participants with only PDA or PFO, without written informed consent, patients older than one year of age or any subject on oxygen at the time of nNO assessment.
  Interventions: Device: Measurement of nasal Nitric Oxide level
- Controls (Active Comparator): The control group will consist of age matched infants, less than one year of age, without CHD or acute respiratory illness. The participants will also require written informed consent and will have to be breathing room air at the time of the nNO test.
  Interventions: Device: Measurement of nasal Nitric Oxide level

INTERVENTIONS:
Device: Measurement of nasal Nitric Oxide level — ECO MEDICS CLD 88 sp Nitric Oxide Analyzer

SUMMARY:
This pilot study aims to measure nasal nitric oxide (nNO) in a group of neonates and infants (≤ 12 months) with congenital heart disease (CHD) and compare their nNO levels to age matched controls without CHD. CHD patients will be divided into subgroups, based on their cardiac anatomy, to try and identify a level of risk of ciliary dyskinesia within the subgroup of CHD. Each of these sub groups' nNO levels will be compared between groups and against age matched control infants without CHD.

DETAILED DESCRIPTION:
Methods: Parents or legal guardians will be approached to provide written, informed consent. To allow for at least three sub groups of cardiac anomalies (with 20 patients per group), 60 children, less than one year of age, with CHD will be recruited from the Pediatric Cardiology inpatient ward at Stollery Children's Hospital. Sixty age matched controls, without acute respiratory illness, will be recruited from the General Pediatric inpatient ward. All subjects will be breathing room air at the time of nNO measurement.

Subjects: This is a pilot study to gather data to power future studies. The investigators aim to recruit 60 subjects with CHD and 60 normal controls without CHD. 60 subjects will allow for at least three sub groups of cardiac anomalies with 20 subjects per group.

Control group: The control group will consist of age matched infants, less than one year of age, without CHD or acute respiratory illness. They will also require written informed consent and will have to be breathing room air at the time of the nNO test.

Investigational device: For nNO assessment, an inert nitric oxide (NO) sampling line with a disposable foam olive (DirectMed Inc., Glen Cove, NY) will be placed into one of the subject's nostrils while the contralateral nostril is left open. Air will be then sampled at a constant rate of 0.3 Liters/min from the nose by a chemiluminescent analyzer which provides measurement of the nNO level in parts per billion (ppb). All nNO measurements will be performed with the subjects supine. Measurements will be obtained using a NO analyzer (CLD 88 SP, ECO PHYSICS AG, Duerten, Switzerland) available at Stollery Children's Hospital. The analyzer will be calibrated according to the manufacturer's specifications. Two samples will be taken five minutes apart, to assess for test-retest reproducibility, with results for each patient being averaged over the two samples. The test is not painful and each sample takes less than a minute.

ELIGIBILITY:
Inclusion Criteria:

* All patients, less than one year of age, with CHD will be eligible for this study with the exception of those patients with only patent foramen ovale (PFO) and patent ductus arteriosus (PDA). The diagnosis of CHD will be confirmed by echocardiography.

Exclusion Criteria:

* All patients, less than one year of age, with CHD will be eligible for this study with the exception of those patients with only patent foramen ovale (PFO) and patent ductus arteriosus (PDA). The diagnosis of CHD will be confirmed by echocardiography.

Control group:

* The control group will consist of age matched infants, less than one year of age, without CHD or acute respiratory illness. They will also require written informed consent and will have to be breathing room air at the time of the nNO test.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2015-12; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
nasal NO level in parts per billion (ppb) | 1 minute

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No